CLINICAL TRIAL: NCT03859427
Title: A Randomized, Open-label, Phase 3 Study Comparing Once-weekly vs Twice-weekly Carfilzomib in Combination With Lenalidomide and Dexamethasone in Subjects With Relapsed or Refractory Multiple Myeloma (A.R.R.O.W.2)
Brief Title: A Study Comparing Once-weekly vs Twice-weekly Carfilzomib in Combination With Lenalidomide and Dexamethasone in Subjects With Relapsed or Refractory Multiple Myeloma
Acronym: ARROW2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180015
Record Dates: First submitted 2019-01-14; First posted 2019-03-01 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: Bone Marrow Cancer
MeSH Terms: conditions — Recurrence; Multiple Myeloma; Bone Marrow Neoplasms | interventions — carfilzomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Carfilzomib once-weekly (Active Comparator): Carfilzomib, lenalidomide, dexamethasone (KRd) regimen using once-weekly carfilzomib 56 mg/m2
  Interventions: Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone
- Carfilzomib twice-weekly (Active Comparator): Carfilzomib, lenalidomide, dexamethasone (KRd) regimen using twice-weekly carfilzomib 27 mg/m2
  Interventions: Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — Once weekly IV over 30 minutes on day 1, 8 and 15 of each 28 day cycle. The dose will be 20 mg/m2 on cycle 1 day 1 and 56 mg/m2 beginning with cycle 1 day 8 and thereafter. 12 cycles or until progression, unacceptable toxicity, death, loss to follow up or withdrawal of consent.
  Arms: Carfilzomib once-weekly
Drug: Carfilzomib — Twice weekly IV over 10 minutes on day 1, 2, 8, 9, 15 and 16 of each 28 day cycle. The dose will be 20 mg/m2 on cycle 1 days 1 and 2 and 27 mg/m2 beginning with cycle 1 day 8 and thereafter. 12 cycles or until progression, unacceptable toxicity, death, loss to follow up or withdrawal of consent.
  Arms: Carfilzomib twice-weekly
Drug: Lenalidomide — Once daily orally 25 mg days 1 to 21 of each cycle. 12 cycles or until progression, unacceptable toxicity, death, loss to follow up or withdrawal of consent
Drug: Dexamethasone — Once daily orally or by IV 40 mg days 1, 8 and 15 of each cycle. Also day 22 of cycles 1 to 9. 12 cycles or until progression, unacceptable toxicity, death, loss to follow up or withdrawal of consent

SUMMARY:
Compare efficacy of 56 mg/m2 carfilzomib administered once-weekly in combination with lenalidomide and dexamethasone (KRd 56 mg/m2) to 27 mg/m2 carfilzomib administered twice-weekly in combination with lenalidomide and dexamethasone (KRd 27 mg/m2) in subjects with relapsed or refractory multiple myeloma (RRMM) with 1 to 3 prior lines of therapy.

ELIGIBILITY:
Inclusion Criteria:

Multiple myeloma with documented relapse or progression after most recent myeloma treatment. Subjects refractory to the most recent line of therapy are eligible, unless last treatment contained proteasome inhibitor (PI) or lenalidomide and dexamethasone. Refractory is defined as disease that is nonresponsive or progresses within 60 days of last therapy.

Subjects must have at least PR to at least 1 line of prior therapy.

Subjects must have received at least 1 but not more than 3 prior lines of therapy for multiple myeloma (induction therapy followed by stem cell transplant and consolidation maintenance therapy will be considered as 1 line of therapy).

Prior therapy with a PI or the combination of lenalidomide and dexamethasone are allowed if the patient had at least a PR to the most recent treatment with a PI or lenalidomide and dexamethasone, neither PI or lenalidomide and dexamethasone containing treatment were ceased due to toxicity, the patient has not relapsed within 60 days of discontinuation of the PI or lenalidomide and dexamethasone containing treatment. A history of prior neuropathy is permitted if this was not grade 3, grade 4 or grade 2 with pain and if not resolved within the 14 days before enrollment, is less than or equal to grade 2 without pain. Patients are permitted to have received single agent lenalidomide as maintenance therapy within 60 days of enrollment.

Previous treatment with a lenalidomide and dexamethasone containing regimen is allowed, as long as the subject did not progress during the first 3 months after initiating lenalidomide and dexamethasone containing therapy.

Measurable disease with at least 1 of the following assessed within 21 days prior to randomization:

* Immunoglobulin G (IgG) multiple myeloma: serum monoclonal protein (M-protein) level ≥ 1.0 g/dL
* Immunoglobulin A (IgA), Immunoglobulin D (IgD), Immunoglobulin E (IgE) multiple myeloma: serum M-protein level ≥ 0.5 g/dL
* Urine M-protein ≥ 200 mg per 24 hours
* In subjects without measurable serum or urine M-protein, serum-free light chain (SFLC) ≥ 100 mg/L (involved light chain) and an abnormal serum kappa lambda ratio

Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 ≤ 2

Other inclusion criteria may apply

Exclusion Criteria:

Waldenström macroglobulinemia.

Multiple myeloma of Immunoglobulin M (IgM) subtype.

Plasma cell leukemia (> 2.0 × 10^9 /L circulating plasma cells by standard differential).

Uncontrolled hypertension, defined as a subject whose blood pressure is greater than or equal to 160 mmHg systolic or greater than or equal to 100 mmHg diastolic when taken in accordance with the European Society of Hypertension/European Society of Cardiology 2018 guidelines (Section 12.10; Williams et al, 2018).

Active congestive heart failure (New York Heart Association Class III to IV), symptomatic ischemia, uncontrolled arrhythmias, screening ECG with corrected QT interval (QTc) of > 470 msec, pericardial disease, or myocardial infarction within 4 months prior to randomization.

Calculated or measured creatinine clearance < 30 mL/min (calculation must be based on the Cockcroft and Gault formula) within 28 days prior to randomization.

Other exclusion criteria may apply

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (108):
- United States (12):
  - Robert A Moss Oncology, Fountain Valley, California
  - Rocky Mountain Cancer Centers Denver Midtown, Denver, Colorado
  - Hartford HealthCare Cancer Institute at The Hospital of Central Connecticut, Plainville, Connecticut
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - New York Oncology Hematology, PC, Albany, New York
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Texas Oncology-Denton, Denton, Texas
  - US Oncology Research Investigational Products Center, Fort Worth, Texas
  - Oncology Consultants PA, Houston, Texas
  - Texas Oncology, San Antonio, Texas
  - United States Oncology Regulatory Affairs Corporate Office, The Woodlands, Texas
- Universitaetsklinikum Salzburg, Salzburg, Austria
- Bulgaria (3):
  - University Multiprofile Hospital for Active Treatment Sveti Georgi EAD, Plovdiv
  - University Multiprofile Hospital for Active Treatment Sveti Ivan Rilski EAD, Sofia
  - Specialized Hospital for Active Treatment of Hematology Diseases EAD, Sofia
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Vseobecna fakultni nemocnice v Praze, Prague
- Finland (3):
  - Helsingin Yliopistollinen Keskussairaala, Helsinki
  - Oulun Yliopistollinen Sairaala, Oulu
  - Turun Yliopistollinen Keskussairaala, Turku
- France (10):
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Centre Hospitalier Universitaire Archet 2, Nice
  - Hopital Saint Louis, Paris
  - Hopital Pitie-Salpetriere, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Poitiers - Hopital la Miletrie, Poitiers
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Institut de Cancerologie Strasbourg, Strasbourg
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
  - Centre Hospitalier Universitaire de Nancy - Hopital de Brabois, Vandœuvre-lès-Nancy
- Germany (5):
  - Charité, Universitätsklinikum Berlin, Campus Benjamin Franklin, Berlin
  - Universitatsklinikum Koln, Cologne
  - Universitätsklinikum Carl Gustav Carus der Technischen Universität Dresden, Dresden
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Johannes Gutenberg Universitaet Mainz, Mainz
- Greece (9):
  - University Hospital of Alexandroupolis, Alexandroupoli
  - General Hospital Evangelismos, Athens
  - Agios Savvas Anticancer Hospital, Athens
  - 251 General Airforce Hospital, Athens
  - Alexandra Hospital, Athens
  - Metropolitan Hospital, Athens
  - General University Hospital of Patras Panagia i Voithia, Pátrai
  - Theagenion Cancer Hospital of Thessaloniki, Thessaloniki
  - General Hospital of Thessaloniki Georgios Papanikolaou, Thessaloniki
- Japan (21):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - Tesshokai Kameda General Hospital, Kamogawa-shi, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Ogaki Municipal Hospital, Ogaki-shi, Gifu
  - National Hospital Organization Shibukawa Medical Center, Shibukawa-shi, Gunma
  - Japanese Red Cross Society Himeji Hospital, Himeji-shi, Hyōgo
  - Hyogo College of Medicine Hospital, Nishinomiya-shi, Hyōgo
  - Hitachi Ltd Hitachi General Hospital, Hitachi-shi, Ibaraki
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - National Hospital Organization Sendai Medical Center, Sendai, Miyagi
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - National Hospital Organization Okayama Medical Center, Okayama, Okayama-ken
  - Japanese Red Cross Osaka Hospital, Osaka, Osaka
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - Saitama Medical Center, Kawagoe-shi, Saitama
  - Tochigi Cancer Center, Utsunomiya, Tochigi
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto-ku, Tokyo
  - Japanese Red Cross Medical Center, Shibuya-ku, Tokyo
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics Public Institution, Kaunas
  - Vilnius University Hospital Santaros Clinic Public Institution, Vilnius
- Netherlands (3):
  - VU Medisch Centrum, Amsterdam
  - Gelre Ziekenhuizen, Apeldoorn
  - Spaarne Gasthuis, Hoofddorp
- Romania (10):
  - Spitalul Clinic Colentina, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Clinic Coltea, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Institutul Oncologic Prof Dr Ion Chiricuta, Cluj-Napoca
  - Institutul Regional de Oncologie Iasi, Iași
  - Spitalul Clinic Dr Gavril Curteanu Oradea, Oradea
  - Spitalul Clinic Judetean de Urgenta Sibiu, Sibiu
  - Spitalul Clinic Municipal de Urgenta Timisoara, Timișoara
- Russia (6):
  - Regional Clinical Hospital, Krasnoyarsk
  - Moscow State Budget Healthcare Institution City clinical Hospital 52 of Moscow Healthcare Department, Moscow
  - SBHI of Moscow city City clinical hospital na S P Botkin of Moscow city Healthcare department, Moscow
  - SBHI of Republic of Karelia Republic Hosiptal n a V A Baranov, Petrozavodsk
  - Federal centre of heart, blood and endocrinology Almazova, Saint Petersburg
  - State Budget Educational Institution of High Professional Skills Samara State Medical University, Samara
- Univerzitna nemocnica Bratislava, Nemocnica sv Cyrila a Metoda, Bratislava, Slovakia
- Spain (6):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Clinico Universitario de Salamanca, Salamanca, Castille and León
  - Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Clinica Universidad de Navarra, Pamplona, Navarre
- Sweden (5):
  - Falu Lasarett, Falun
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Hallands Sjukhus Halmstad, Halmstad
  - Sunderby Sjukhus, Luleå
  - Skanes Universitetssjukhus, Lund
- Turkey (Türkiye) (7):
  - Gazi Universitesi Saglik Arastirma ve Uygulama Merkezi Gazi Hastanesi, Ankara
  - Ankara Universitesi Tip Fakultesi Cebeci Arastirma ve Uygulama Hastanesi, Ankara
  - Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul
  - Bagcilar Medipol Mega Universite Hastanesi, Istanbul
  - Istanbul Florence Nightingale Hastanesi, Istanbul
  - Dokuz Eylul Universitesi Arastirma Uygulama Hastanesi, Izmir
  - Erciyes Universitesi Tip Fakultesi Mehmet Kemal Dedeman Hematoloji-Onkoloji Hastanesi, Kayseri

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Dimopoulos MA, Coriu D, Delimpasi S, Spicka I, Upchurch T, Fang B, Talpur R, Faber E, Beksac M, Leleu X. A.R.R.O.W.2: once- vs twice-weekly carfilzomib, lenalidomide, and dexamethasone in relapsed/refractory multiple myeloma. Blood Adv. 2024 Oct 8;8(19):5012-5021. doi: 10.1182/bloodadvances.2024013101. PMID 39024542
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 80 study centers in Europe, Japan, and the United States, and participated from 08 May 2019 to 31 March 2023.
Pre-assignment Details: Participants with relapsed or refractory multiple myeloma were randomized in a 1:1 ratio to receive once-weekly or twice-weekly carfilzomib. Randomization was stratified by original International Staging System (ISS) stage at the time of study entry (stage 1 or 2 versus stage 3), prior lenalidomide treatment (yes versus no), prior proteasome inhibitor treatment (yes versus no), and prior anti-CD38 exposure (yes versus no).
Groups:
- Twice-weekly Kyprolis (Carfilzomib) + Lenalidomide + Dexamethsone (KRd) 20/27 mg/m^2: Carfilzomib was administered twice-weekly intravenously as a 10 ± 5 minute infusion using an infusion pump on Days 1, 2, 8, 9, 15, and 16 of each 28-day cycle. The dose was 20 mg/m^2 on Days 1 and 2 of Cycle 1 and 27 mg/m^2 beginning on Day 8 of Cycle 1 and thereafter. Participants also received lenalidomide 25 mg daily orally on Days 1 to 21 of each cycle and dexamethasone 40 mg weekly orally or intravenously. Participants were treated for up to 12 28-day cycles.
- Once-weekly KRd 20/56 mg/m^2: Carfilzomib was administered once-weekly intravenously as a 30 ± 5 minute infusion using an infusion pump on Days 1, 8, and 15 of each 28-day cycle. The dose was 20 mg/m^2 on Day 1 of Cycle 1 and 56 mg/m^2 beginning on Day 8 of Cycle 1 and thereafter. Participants also received lenalidomide 25 mg daily orally on Days 1 to 21 of each cycle and dexamethasone 40 mg weekly orally or intravenously. Participants were treated for up to 12 28-day cycles.
Period: Overall Study
Arm/Group | Twice-weekly Kyprolis (Carfilzomib) + Lenalidomide + Dexamethsone (KRd) 20/27 mg/m^2 | Once-weekly KRd 20/56 mg/m^2
Started | 226 | 228
Received Carfilzomib | 226 | 228
Completed 12 Cycles Carfilzomib | 152 | 150
Received Lenalidomide | 226 | 228
Received Dexamethasone | 226 | 228
Safety Population (Participants were analyzed according to the treatment arm corresponding to the actual treatment received.) | 231 | 223
Completed | 197 | 191
Not Completed | 29 | 37
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Decision by sponsor | 0 | 3
Not completed — Lost to Follow-up | 3 | 2
Not completed — Death | 22 | 25

BASELINE CHARACTERISTICS:
Groups:
- Twice-weekly KRd 20/27 mg/m^2: Carfilzomib was administered twice-weekly intravenously as a 10 ± 5 minute infusion using an infusion pump on Days 1, 2, 8, 9, 15, and 16 of each 28-day cycle. The dose was 20 mg/m^2 on Days 1 and 2 of Cycle 1 and 27 mg/m^2 beginning on Day 8 of Cycle 1 and thereafter. Participants also received lenalidomide 25 mg daily orally on Days 1 to 21 of each cycle and dexamethasone 40 mg weekly orally or intravenously. Participants were treated for up to 12 28-day cycles.
- Total: Total of all reporting groups
Arm/Group | Twice-weekly KRd 20/27 mg/m^2 | Once-weekly KRd 20/56 mg/m^2 | Total
Number analyzed (Participants) | 226 | 228 | 454
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (8.2) | 63.7 (8.4) | 63.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 118 | 218
  Male | 126 | 110 | 236
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 213 | 215 | 428
  Unknown or Not Reported | 5 | 5 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 12 | 21
  Black or African American | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 209 | 209 | 418
  Other | 7 | 6 | 13
Original ISS Stage at Study Entry [Count of Participants; unit: Participants] — ISS stage classification at study entry per interactive voice/web response system for randomization. Stage 1: serum beta-2 microglobulin < 3.5 mg/L and serum albumin ≥ 3.5 g/dL; Stage 2: serum beta-2 microglobulin < 3.5 mg/L and serum albumin < 3.5 g/dL or serum beta-2 microglobulin 3.5 - < 5.5 mg/L irrespective of the serum albumin; Stage 3: serum beta-2 microglobulin ≥ 5.5 mg/L.
  Participants
    Stage 1 or 2 | 201 | 201 | 402
    Stage 3 | 25 | 27 | 52
Prior Lenalidomide Treatment [Count of Participants; unit: Participants]
  Yes | 79 | 85 | 164
  No | 147 | 143 | 290
Prior Proteasome Inhibitor Treatment [Count of Participants; unit: Participants]
  Yes | 218 | 214 | 432
  No | 8 | 14 | 22
Prior Anti-CD38 Treatment [Count of Participants; unit: Participants]
  Yes | 17 | 21 | 38
  No | 209 | 207 | 416

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Per International Myeloma Working Group Uniform Response Criteria (IMWG-URC)
Description: ORR was defined as the percentage of participants with a best overall response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) per IMWG-URC. CR: negative immunofixation on serum and urine, soft tissue plasmacytomas disappearance, < 5% plasma cells in bone marrow (BM). sCR: CR and normal serum free light chain ratio and no clonal cells in BM by immunohistochemistry. VGPR: Serum and urine M-protein detectable by immunofixation or ≥ 90% reduction in serum M-protein (urine M-protein level < 100 mg/24-hours). PR: ≥ 50% reduction of serum M-protein and reduction in 24-hours urinary M-protein by ≥ 90% or to < 200 mg/24-hours. The ORR 95% confidence intervals (CIs) were estimated using the Clopper-Pearson method.
Time Frame: Cycle 1 Day 1 up to approximately 12 months (cycle = 28 days); median treatment duration for the twice-weekly arm was 47.00 weeks and for the once-weekly arm was 47.14 weeks.
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Twice-weekly KRd 20/27 mg/m^2 | Once-weekly KRd 20/56 mg/m^2
Number analyzed (Participants) | 226 | 228
percentage of participants | 86.3 [81.1 to 90.5] | 82.5 [76.9 to 87.2]
Statistical Analysis 1: Comparison: Twice-weekly KRd 20/27 mg/m^2 vs Once-weekly KRd 20/56 mg/m^2; Test type: Non-Inferiority — The non-inferiority margin was 0.87 for the estimated ORR risk ratio; p = 0.0666, Synthesis approach — P-value (2.5% significance level) of the non-inferiority test via the synthesis approach (FDA, 2016) for non-inferiority comparison of ORR between treatment arms; Risk Ratio (RR) = 0.954, 95% CI 2-sided [0.882 to 1.032] — Risk ratio and 95% CIs were estimated by a stratified analysis using the Cochran-Mantel-Haenszel method

2. Secondary Outcome: Kaplan-Meier Estimate of Progression-free Survival (PFS) Rate at 12 Months
Description: PFS rate was defined as the percentage of participants without disease progression or death due to any cause at 12 months. The PFS rate at 12 months was estimated using the Kaplan-Meier method by Klein and Moeschberger (1997). 95% CIs were estimated using the method by Kalbfleisch and Prentice (1980). PFS data was censored for participants who met any one of the following: 1. no baseline/no post-baseline disease assessments; 2. starting new anti-myeloma therapy before documentation of progressive disease (PD) or death; 3. PD or death immediately after more than 1 consecutively missed disease assessment visit (PD or death immediately after > 63 days without disease assessment visit); 4. alive without documentation of PD; 5. lost to follow-up or withdrawn consent.
Time Frame: 12 months
Population: The ITT analysis set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Twice-weekly KRd 20/27 mg/m^2 | Once-weekly KRd 20/56 mg/m^2
Number analyzed (Participants) | 226 | 228
percentage of participants | 79.7 [73.6 to 84.6] | 80.7 [74.7 to 85.4]

3. Secondary Outcome: Percentage of Participants Who Reported Convenience as Measured by the Patient-reported Convenience With Carfilzomib-dosing Schedule Question
Description: Patient-reported convenience was measured by the Patient-reported Convenience with Carfilzomib-dosing Schedule Question. The items in the questionnaire were categorized as 'Convenient', which included responses of 'Very Convenient' and 'Convenient', and 'Inconvenient' which included responses of 'Inconvenient' and 'Very Inconvenient'. The 95% CIs were estimated using the Clopper-Pearson method.
Time Frame: Day 28 of Cycle 4
Population: The ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Twice-weekly KRd 20/27 mg/m^2 | Once-weekly KRd 20/56 mg/m^2
Number analyzed (Participants) | 226 | 228
percentage of participants | 80.5 [74.8 to 85.5] | 81.6 [75.9 to 86.4]
Statistical Analysis 1: Comparison: Twice-weekly KRd 20/27 mg/m^2 vs Once-weekly KRd 20/56 mg/m^2; Test type: Other; Odds Ratio (OR) = 1.049, 95% CI 2-sided [0.653 to 1.683] — Odds ratio and 95% CIs were estimated by a stratified analysis using the Cochran-Mantel-Haenszel method

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment. TEAEs were AEs starting on or after the first dose of any study drug, and up to 30 days of the last dose of any study drug, excluding AEs reported after End of Study date.
Time Frame: Cycle 1 Day 1 up to end of Cycle 12 + 30 days, where each cycle was 28 days; median treatment duration (any study treatment) was 47.00 weeks in the twice-weekly KRd group and 47.14 weeks in the once-weekly KRd group
Population: The safety population included all randomized participants who received at least 1 dose of any study treatment (carfilzomib, lenalidomide, or dexamethasone). Participants were analyzed according to the treatment arm corresponding to the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Twice-weekly KRd 20/27 mg/m^2 | Once-weekly KRd 20/56 mg/m^2
Number analyzed (Participants) | 231 | 223
Participants | 219 | 209

5. Secondary Outcome: Time to Response (TTR)
Description: TTR was defined as the time from randomization to the earliest date when confirmed sCR, CR, VGPR, or PR per IMWG-URC was first achieved.
Time Frame: as for outcome 1
Population: The ITT population included all randomized participants. Data is presented for participants in the ITT population who achieved a confirmed response of PR or better.
Measure: Median (Full Range); unit: months
Arm/Group | Twice-weekly KRd 20/27 mg/m^2 | Once-weekly KRd 20/56 mg/m^2
Number analyzed (Participants) | 195 | 188
months | 1.0 [1 to 12] | 1.0 [1 to 10]

6. Secondary Outcome: Kaplan-Meier Estimate of Duration of Response (DOR)
Description: For participants who achieved a PR or better, i.e., sCR, CR, VGPR, or PR per IMWG-URC, the DOR was defined as the time from the earliest date when a PR or better was first achieved, and subsequently confirmed, to the earliest date of confirmed PD or death due to any cause. Median DOR was estimated using the Kaplan-Meier method. 95% CIs were estimated using the method by Klein and Moeschberger (1997) with log-log transformation. For those alive and who had not experienced PD by analysis time, DOR was censored for participants who met any one of the following: 1. no baseline/no post-baseline disease assessments; 2. starting new anti-myeloma therapy before documentation of PD or death; 3. PD or death immediately after more than 1 consecutively missed disease assessment visit (PD or death immediately after > 63 days without disease assessment visit); 4. alive without documentation of PD; 5. lost to follow-up or withdrawn consent.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Median (Full Range); unit: months
Arm/Group | Twice-weekly KRd 20/27 mg/m^2 | Once-weekly KRd 20/56 mg/m^2
Number analyzed (Participants) | 195 | 188
months | NA [NA to NA] — The median and 95% CIs could not be estimated due to too few events. | NA [NA to NA] — The median and 95% CIs could not be estimated due to too few events.

7. Secondary Outcome: Kaplan-Meier Estimate of Time to Progression (TTP)
Description: TTP was defined as the duration from randomization for the first documented disease progression per IMWG-UCR. Median TTP was estimated using the Kaplan-Meier method. 95% CIs were estimated using the method by Klein and Moeschberger (1997) with log-log transformation. TTP was censored for participants who had no confirmed PD at the last non non-evaluable (non-NE), post-baseline disease assessment or the earlier of the following, where applicable: 1. the last non-NE, post-baseline disease assessment prior to start of a new anti-myeloma treatment, or 2. the last non-NE, post-baseline assessment followed > 63 days later by disease progression; otherwise, at randomization.
Time Frame: as for outcome 1
Population: The ITT population included all randomized participants.
Measure: Median (Full Range); unit: months
Arm/Group | Twice-weekly KRd 20/27 mg/m^2 | Once-weekly KRd 20/56 mg/m^2
Number analyzed (Participants) | 226 | 228
months | NA [NA to NA] — The median and 95% CIs could not be estimated due to too few events. | NA [NA to NA] — The median and 95% CIs could not be estimated due to too few events.

8. Secondary Outcome: Kaplan-Meier Estimate of Overall Survival (OS)
Description: OS was defined as the time from randomization to the date of death due to any cause. Median OS was estimated using the Kaplan-Meier method. 95% CIs were estimated using the method by Klein and Moeschberger (1997) with log-log transformation. Participants still alive or lost to follow-up or withdrawn consent from study by the analysis time were censored at the date on which the participant was last known to be alive.
Time Frame: as for outcome 1
Population: The ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Twice-weekly KRd 20/27 mg/m^2 | Once-weekly KRd 20/56 mg/m^2
Number analyzed (Participants) | 226 | 228
months | NA [NA to NA] — The median and 95% CIs could not be estimated due to too few events. | NA [NA to NA] — The median and 95% CIs could not be estimated due to too few events.

9. Secondary Outcome: Percentage of Participants Who Achieved Minimal Residual Disease Negative Complete Response (MRD[-]CR) by Independent Review Committee (IRC) Per IMWG-URC
Description: MRD[-]CR was defined as achievement of CR or better by IRC per IMWG-URC and achievement of MRD negativity as assessed by next generation sequencing method at a 10^-5 threshold over the duration of the study. The 95% CIs for percentages were estimated using the Clopper-Pearson method.
Time Frame: as for outcome 1
Population: The ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Twice-weekly KRd 20/27 mg/m^2 | Once-weekly KRd 20/56 mg/m^2
Number analyzed (Participants) | 226 | 228
percentage of participants | 18.1 [13.3 to 23.8] | 21.5 [16.3 to 27.4]
Statistical Analysis 1: Comparison: Twice-weekly KRd 20/27 mg/m^2 vs Once-weekly KRd 20/56 mg/m^2; Test type: Other; Odds Ratio (OR) = 1.235, 95% CI 2-sided [0.775 to 1.970] — Odds ratio and 95% CIs were estimated by a stratified analysis using the Cochran-Mantel-Haenszel method

10. Secondary Outcome: Percentage of Participants With Minimal Residual Disease Negativity (MRD[-]) by IRC Per IMWG-URC at 12 Months
Description: The percentage of participants with achievement of MRD[-] at 12 months (± 4 weeks) from randomization, as assessed by next generation sequencing method at a 10^-5 threshold. MRD negativity results from BM samples obtained at 8 to 13 months from randomization and prior to new anti-myeloma therapy or disease progression were considered in the calculation. The 95% CIs for percentages were estimated using the Clopper-Pearson method.
Time Frame: Cycle 1 Day 1 up to 12 months (cycle = 28 days)
Population: The ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Twice-weekly KRd 20/27 mg/m^2 | Once-weekly KRd 20/56 mg/m^2
Number analyzed (Participants) | 226 | 228
percentage of participants | 18.1 [13.3 to 23.8] | 18.9 [14.0 to 24.6]
Statistical Analysis 1: Comparison: Twice-weekly KRd 20/27 mg/m^2 vs Once-weekly KRd 20/56 mg/m^2; Test type: Other; Odds Ratio (OR) = 1.060, 95% CI 2-sided [0.657 to 1.711] — Odds ratio and 95% CIs were estimated by a stratified analysis using the Cochran-Mantel-Haenszel method

11. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire (EORTC QLQ)-Core 30 (C30) Physical Functioning Scale
Description: The QLQ-C30 physical function is one of the functional domains of the EORTC QLQ-C30 self-reported instrument and the physical functioning score score ranges from 0-100 points, with 100 points indicating the best possible functioning. A positive change from baseline indicated an improvement in functioning.
Time Frame: Baseline (Cycle 1 Day 1), Cycle 3 Day 1, Cycle 5 Day 1, Cycle 7 Day 1, Cycle 9 Day 1, Cycle 12 Day 1, and safety follow-up (30 days after last dose)
Population: The ITT population included all randomized participants. Participants with data available at each time point are presented. All participants in the overall number of participants analyzed contributed to the data in the endpoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Twice-weekly KRd 20/27 mg/m^2 | Once-weekly KRd 20/56 mg/m^2
Number analyzed (Participants) | 226 | 228
Score on a scale
  Cycle 3 Day 1: number analyzed (Participants) | 186 | 182
  Cycle 3 Day 1 | -2.76 (16.84) | -0.77 (14.95)
  Cycle 5 Day 1: number analyzed (Participants) | 181 | 177
  Cycle 5 Day 1 | -2.65 (15.76) | 0.26 (15.59)
  Cycle 7 Day 1: number analyzed (Participants) | 162 | 161
  Cycle 7 Day 1 | -0.82 (16.59) | 0.17 (14.62)
  Cycle 9 Day 1: number analyzed (Participants) | 152 | 148
  Cycle 9 Day 1 | -1.05 (15.59) | 2.03 (14.75)
  Cycle 12 Day 1: number analyzed (Participants) | 134 | 132
  Cycle 12 Day 1 | -1.89 (15.15) | 1.06 (15.63)
  Safety Follow-up: number analyzed (Participants) | 146 | 145
  Safety Follow-up | -1.55 (16.31) | 2.11 (18.27)
Statistical Analysis 1: Comparison: Twice-weekly KRd 20/27 mg/m^2 vs Once-weekly KRd 20/56 mg/m^2; Test type: Other; Least Squares (LS) Mean Difference = 2.53, 95% CI 2-sided [0.38 to 4.69] — Analysis was based on repeated measures analysis of covariance (ANCOVA) model, including arm, baseline scale score, randomization stratification factors and visit as repeated measure

12. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 Role Functioning Scale
Description: The QLQ-C30 role function is one of the functional domains of the EORTC QLQ-C30 self-reported instrument and the role functioning score ranges from 0-100 points, with 100 points indicating the best possible functioning. A positive change from baseline indicated an improvement in functioning.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Twice-weekly KRd 20/27 mg/m^2 | Once-weekly KRd 20/56 mg/m^2
Number analyzed (Participants) | 226 | 228
Score on a scale
  Cycle 3 Day 1: number analyzed (Participants) | 186 | 182
  Cycle 3 Day 1 | -4.30 (26.16) | -2.47 (24.81)
  Cycle 5 Day 1: number analyzed (Participants) | 181 | 177
  Cycle 5 Day 1 | -2.67 (25.77) | -3.11 (24.32)
  Cycle 7 Day 1: number analyzed (Participants) | 162 | 161
  Cycle 7 Day 1 | -3.29 (26.19) | 1.76 (24.34)
  Cycle 9 Day 1: number analyzed (Participants) | 152 | 148
  Cycle 9 Day 1 | -0.88 (23.24) | 2.70 (24.90)
  Cycle 12 Day 1: number analyzed (Participants) | 134 | 132
  Cycle 12 Day 1 | -0.25 (23.21) | 1.64 (28.97)
  Safety Follow-up: number analyzed (Participants) | 146 | 145
  Safety Follow-up | -2.28 (24.73) | 3.68 (26.24)
Statistical Analysis 1: Comparison: Twice-weekly KRd 20/27 mg/m^2 vs Once-weekly KRd 20/56 mg/m^2; Test type: Other; LS Mean Difference = 1.73, 95% CI 2-sided [-1.26 to 4.72] — Analysis was based on ANCOVA model, including arm, baseline scale score, randomization stratification factors and visit as repeated measure

13. Secondary Outcome: Patient-reported Treatment Satisfaction as Measured by the Cancer Therapy Satisfaction Questionnaire (CTSQ)
Description: The CTSQ measures treatment satisfaction in individuals with cancer and includes a domain for satisfaction with therapy. The satisfaction with therapy scores ranges from 0 to 100 points, with 100 points indicating greatest satisfaction.
  Analysis was based on ANCOVA model. The dependent variable of the models were the scale scores measured at each visit. The model included effects of intercept, scale score measured at cycle 2 day 1 visit, treatment arm, and randomization stratification factors.
Time Frame: Cycle 5 Day 1, Cycle 12 Day 1, and safety follow-up (30 days after last dose)
Population: The ITT population included all randomized participants. Participants with data available at each time point are presented.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Twice-weekly KRd 20/27 mg/m^2 | Once-weekly KRd 20/56 mg/m^2
Number analyzed (Participants) | 169 | 165
Score on a scale
  Cycle 5 Day 1 | 75.73 (1.78) | 75.47 (1.76)
  Cycle 12 Day 1: number analyzed (Participants) | 128 | 122
  Cycle 12 Day 1 | 78.39 (2.40) | 77.91 (2.40)
  Safety follow-up: number analyzed (Participants) | 138 | 134
  Safety follow-up | 74.55 (2.58) | 75.99 (2.49)
Statistical Analysis 1: Comparison: Twice-weekly KRd 20/27 mg/m^2 vs Once-weekly KRd 20/56 mg/m^2; Test type: Other; LS Mean difference = -0.26, 95% CI 2-sided [-2.54 to 2.03], Standard Error of Mean 1.16 — Treatment difference at Cycle 5
Statistical Analysis 2: Comparison: Twice-weekly KRd 20/27 mg/m^2 vs Once-weekly KRd 20/56 mg/m^2; Test type: Other; LS Mean difference = -0.48, 95% CI 2-sided [-3.24 to 2.28], Standard Error of Mean 1.40 — Treatment difference at Cycle 12
Statistical Analysis 3: Comparison: Twice-weekly KRd 20/27 mg/m^2 vs Once-weekly KRd 20/56 mg/m^2; Test type: Other; LS Mean difference = 1.44, 95% CI 2-sided [-1.69 to 4.58], Standard Error of Mean 1.59 — Treatment difference at safety follow-up

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected from enrollment to End of Study; median study duration was 12.0 months. AEs were collected from first dose of study drug to last dose of study drug + 30 days; median treatment duration (any study treatment) was 11.8 months.
Description: All-cause mortality was collected for all participants enrolled/randomized in the study and is presented according to the randomized treatment arm. Serious AEs and other AEs were collected for all participants in the safety population who received at least one dose of study drug. Participants in the safety population were analyzed according to the treatment arm corresponding to the actual treatment received.
Arm/Group | Twice-weekly KRd 20/27 mg/m^2 | Once-weekly KRd 20/56 mg/m^2
All-Cause Mortality (participants affected / at risk) | 22/226 | 26/228
Serious Adverse Events (participants affected / at risk) | 75/231 | 84/223
Other Adverse Events (participants affected / at risk) | 190/231 | 182/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Twice-weekly KRd 20/27 mg/m^2 (N=231) | Once-weekly KRd 20/56 mg/m^2 (N=223)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Death (General disorders) | 0 | 3
General physical health deterioration (General disorders) | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 2
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
COVID-19 (Infections and infestations) | 3 | 6
COVID-19 pneumonia (Infections and infestations) | 11 | 8
Coronavirus infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 2
Influenza (Infections and infestations) | 2 | 1
Intervertebral discitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 9 | 12
Pneumonia bacterial (Infections and infestations) | 0 | 2
Pneumonia haemophilus (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 3
Septic shock (Infections and infestations) | 0 | 1
Sinobronchitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Superinfection bacterial (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 2
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Electrocardiogram abnormal (Investigations) | 1 | 0
Hepatic enzyme abnormal (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Amplified musculoskeletal pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 0 | 1
Intensive care unit acquired weakness (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 1
Lacunar stroke (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Cryoglobulinaemia (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 2
Peripheral venous disease (Vascular disorders) | 1 | 0
Poor venous access (Vascular disorders) | 1 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Twice-weekly KRd 20/27 mg/m^2 (N=231) | Once-weekly KRd 20/56 mg/m^2 (N=223)
Anaemia (Blood and lymphatic system disorders) | 55 | 56
Neutropenia (Blood and lymphatic system disorders) | 73 | 65
Thrombocytopenia (Blood and lymphatic system disorders) | 31 | 46
Constipation (Gastrointestinal disorders) | 17 | 23
Diarrhoea (Gastrointestinal disorders) | 43 | 42
Nausea (Gastrointestinal disorders) | 15 | 19
Asthenia (General disorders) | 13 | 26
Fatigue (General disorders) | 29 | 24
Pyrexia (General disorders) | 27 | 23
Hepatic function abnormal (Hepatobiliary disorders) | 8 | 12
Bronchitis (Infections and infestations) | 15 | 11
COVID-19 (Infections and infestations) | 14 | 22
Nasopharyngitis (Infections and infestations) | 16 | 16
Upper respiratory tract infection (Infections and infestations) | 33 | 32
Hyperglycaemia (Metabolism and nutrition disorders) | 17 | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 13 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 18 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 17
Muscle spasms (Musculoskeletal and connective tissue disorders) | 21 | 12
Headache (Nervous system disorders) | 12 | 9
Neuropathy peripheral (Nervous system disorders) | 11 | 22
Insomnia (Psychiatric disorders) | 16 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 13
Rash (Skin and subcutaneous tissue disorders) | 16 | 21
Hypertension (Vascular disorders) | 56 | 48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT03859427/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT03859427/SAP_001.pdf